CLINICAL TRIAL: NCT01541761
Title: RCT Testing the Effectiveness of an Early Obesity Prevention Program
Brief Title: Starting Early Obesity Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-02175
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Childhood Obesity
Keywords: Obesity; Child; Hispanic; Prevention; Nutrition; Parenting
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family groups (Experimental): Intervention group members will participate in family groups focused on early childhood obesity prevention in addition to standard care from pediatricians at the primary care clinic.
  Interventions: Behavioral: Family groups
- Standard care (No Intervention): Mothers enrolled into the control group will continue to receive care from their pediatrician in the primary care clinic.

INTERVENTIONS:
Behavioral: Family groups — The group sessions are designed to facilitate on-going interaction among consistent groups of 6 - 8 parents and other care givers with infants the same age and will be coordinated with scheduled well child care visits. They will be conducted in English and Spanish. The groups will focus on nutrition and, parenting.
  Arms: Family groups

SUMMARY:
The proposed study is a randomized controlled trial to test the effectiveness of a primary care, family-centered child obesity prevention program beginning in pregnancy and continuing throughout the first three years of life compared to routine standard of care. The study aims to reduce the prevalence of obesity at age three, improve child diet composition and healthy lifestyle behaviors. Pregnant women will be enrolled from a large urban medical center serving primarily low-income immigrant Latino families. The intervention "Starting Early" will consist of three components. 1) Family Groups: interactive groups coordinated with the child's primary care visits and led by a Nutritionist/ Child Developmental Specialist. 2) Nutritional Video: a culturally-specific bilingual early nutrition video will be incorporated into family group discussions. 3) Plain Language Handouts: given to reinforce the curriculum from the family groups.

The proposed research included in the funding continuation is titled: "Starting Early: Expansion of a Primary Care-Based Early Child Obesity Prevention Program". It adds three major components to the current project: 1) Following the original Starting Early cohort until age 5; 2) Developing and piloting an extended Starting Early preschool intervention for children aged 3-5 years.; 3) Developing and piloting an extended Starting Early prenatal intervention for women in the 1st trimester of pregnancy. A new cohort of 200 women in the first trimester of pregnancy will be recruited for the prenatal intervention; all women will receive the intervention in this feasibility trial.

Hypothesis: Compared to controls, the intervention group will show reduced obesity and improved parent feeding knowledge and increased healthy feeding attitudes, styles and practices

DETAILED DESCRIPTION:
Expected outcomes include: (1) Reduction in the prevalence and degree of obesity. (2) Improvement in child diet composition. (3) Improvement in parent feeding knowledge, attitudes, styles and practices including. (4) Improvement in lifestyle behaviors, such as sleep, screen time and physical activity, associated with increased risk of obesity. (5) Improvement in parent diet.

Our secondary objective is to understand the mechanisms by which changes in parent knowledge and behavioral factors mediate impacts of the intervention on childhood obesity. We will also study relationships between potential moderators and intervention impacts. The new components of the expanded Starting Early Program will be feasible: Families will participate in the preschool intervention, and pregnant women will enroll in the prenatal intervention.

ELIGIBILITY:
Inclusion Criteria:

* Latina mother > 18 years with singleton uncomplicated pregnancy
* Receiving prenatal care and the intention to receive pediatric care at Bellevue Hospital Center or Gouverneur Healthcare Services
* Mother to be primary caregiver of child
* Mother speaks fluent English or Spanish

Exclusion Criteria:

* Maternal history of serious medical or psychiatric illness or drug or alcohol abuse
* Family does not have a phone
* Infants with severe medical problems that may affect feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Reduction in the prevalence and degree of obesity at age 3 years | 3 years
  Continuous and dichotomized measures (BMI percentiles)
Improvement in infant diet composition | 1-3 years
  Diets of intervention group infants and children will be more likely to follow recommended guidelines including:
  i) Increased breastfeeding rates and duration ii) Appropriate timing of introduction to solids iii) Appropriate timing of bottle weaning iv) Increased fruit and vegetable consumption v) Decreased fast and junk food consumption vi) Decreased sugary beverage consumption vii) Age-appropriate portion sizes
Improvement in infant lifestyle behaviors associated with increased risk of obesity. | 1-3 years
  Measures of lifestyle behaviors among infants and children receiving intervention will be more likely to follow recommended guidelines than those of the control group including:
  i) Better sleep habits ii) Reduced screen time iii) Increased physical activity
Improvement in parent feeding knowledge, attitudes, styles and practices | 1-3 years
  Parent feeding knowledge, attitudes, styles and practices in the intervention group will be healthier than those of the control group including:
  i) Awareness of healthy child weight ii) Improved knowledge of optimal feeding practices iii) More responsive feeding style
Reduction in infant and child excess weight gain | 1-3 years
  Continuous anthropometric measures (weight for length z-scores)
Additional Outcome Measures for the Expanded Starting Early Program: Preschool intervention | 2-5 years
  Will be feasible, intervention mothers will have improved nutrition knowledge, and feeding attitudes, styles and behaviors
Additional Outcome Measures for the Expanded Starting Early Program: Prenatal Intervention | 2-5 years
  Will be feasible, ii) intervention women will have improved nutrition knowledge and behaviors, iii) intervention women will have improved gestational weight gain
Feasibility process measures: | 2-5 years
  Study population eligibility and enrollment, Proportion of pregnant women approached who meet eligibility criteria, Proportion of women meeting eligibility criteria who enroll These proportions will be calculated using study recruitment records.
Participant engagement | 2-5 years
  Proportion of enrolled mother-infant dyads that participate in the different aspects of the program. This will include the number of individual sessions with healthy steps, the number of individual sessions with the health educator, the number and type of referrals to community resources provided, and the number of Nutrition and Parenting Support Groups attended. This will enable us to determine the length of engagement in the program, proportion of enrolled mother-infant dyads that complete each study measure
Participant satisfaction | 2-5 years
  We will assess program satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Messito, MD, Principal Investigator — NYU School of Medicine; Rachel Gross, MD MS, Principal Investigator — Children's Hospital at Montefiore
Locations (1):
- Bellevue Hospital Center Ambulatory Care Clinic, New York, New York, United States

REFERENCES:
- [Derived] Duh-Leong C, Messito MJ, Katzow MW, Kim CN, Mendelsohn AL, Scott MA, Gross RS. Prenatal and Pediatric Primary Care-Based Child Obesity Prevention: Effects of Adverse Social Determinants of Health on Intervention Attendance and Impact. Child Obes. 2024 Oct;20(7):476-484. doi: 10.1089/chi.2023.0149. Epub 2024 Feb 1. PMID 38301173
- [Derived] Vandyousefi S, Messito MJ, Scott MA, Gross RS. Do Appetite Traits Mediate the Link Between Birth Weight and Later Child Weight in Low-Income Hispanic Families? Child Obes. 2023 Oct;19(7):489-497. doi: 10.1089/chi.2022.0124. Epub 2022 Oct 17. PMID 36255444
- [Derived] Katzow MW, Messito MJ, Mendelsohn AL, Scott MA, Gross RS. Protective Effect of Prenatal Social Support on the Intergenerational Transmission of Obesity in Low-Income Hispanic Families. Child Obes. 2023 Sep;19(6):382-390. doi: 10.1089/chi.2021.0306. Epub 2022 Sep 15. PMID 36112108
- [Derived] Messito MJ, Mendelsohn AL, Katzow MW, Scott MA, Vandyousefi S, Gross RS. Prenatal and Pediatric Primary Care-Based Child Obesity Prevention Program: A Randomized Trial. Pediatrics. 2020 Oct;146(4):e20200709. doi: 10.1542/peds.2020-0709. Epub 2020 Sep 3. PMID 32883807
- [Derived] Gross RS, Mendelsohn AL, Yin HS, Tomopoulos S, Gross MB, Scheinmann R, Messito MJ. Randomized controlled trial of an early child obesity prevention intervention: Impacts on infant tummy time. Obesity (Silver Spring). 2017 May;25(5):920-927. doi: 10.1002/oby.21779. Epub 2017 Mar 22. PMID 28332324
- [Derived] Gross RS, Mendelsohn AL, Gross MB, Scheinmann R, Messito MJ. Randomized Controlled Trial of a Primary Care-Based Child Obesity Prevention Intervention on Infant Feeding Practices. J Pediatr. 2016 Jul;174:171-177.e2. doi: 10.1016/j.jpeds.2016.03.060. Epub 2016 Apr 21. PMID 27113376